CLINICAL TRIAL: NCT06917222
Title: Slide Tracheoplasty Versus Tracheal Resection Anastomosis in Acquired Tracheal Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Eslam Hamed Elsayed Abdou, Assistant lecturer, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Slide tracheoplasty
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-04

CONDITIONS: Tracheal Stenosis; Subglottic Stenosis
Keywords: Slide tracheoplasty; Tracheal resection anastomosis
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slide tracheoplasty (Experimental)
  Interventions: Procedure: Slide tracheoplasty
- Tracheal resection anastomosis (Experimental)
  Interventions: Procedure: Tracheal resection anastomosis

INTERVENTIONS:
Procedure: Slide tracheoplasty — Management of tracheal stenosis by slide tracheoplasty
  Arms: Slide tracheoplasty
Procedure: Tracheal resection anastomosis — Management of tracheal stenosis by tracheal resection anastomosis
  Arms: Tracheal resection anastomosis

SUMMARY:
Aim of the Work To compare the clinical outcomes between patients will undergo slide tracheoplasty and those will undergo tracheal resection anastomosis for acquired tracheal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with grade III, IV acquired tracheal stenosis (e.g., due to trauma, prolonged intubation) regardless their age or sex.

  * Patient with symptomatic high grade II acquired laryngotracheal stenosis after failure of endoscopic interventions.
  * Clinical indications for surgical intervention (Symptoms of airway obstruction).
  * Feasible for surgical intervention.

Exclusion Criteria:

* congenital tracheal stenosis

  * Malignant stenosis.
  * Severe comorbidities that contraindicate the surgery.
  * Patients refusing to sign the consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Success Rate of Procedure | 3-6 months
  Defined as the absence of stridor or the need for re-intervention within a defined follow-up period (3 months

SECONDARY OUTCOMES:
Complication Rates | 3 months
  Evaluation of perioperative complications:
  * Immediate Complications: Airway obstruction, pneumothorax, anastomotic leak, or accidental injury to surrounding structures (e.g., RLN).
  * Delayed Complications: Stenosis, granulation tissue formation, tracheomalacia, or infection (e.g., mediastinitis).
  * Mortality Rate: Intraoperative and 30-day mortality rates
Duration of Hospital Stay | 3 months
  Measured from the day of surgery to discharge
Time to Decannulation | 3 months
  Time taken for patients to be successfully decannulated, which can be indicative of recovery and airway stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Eslam Hamed, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bocage JP, Caccavale R, Lewis R, Sisler G, MacKenzie J. Tracheal stenosis. N J Med. 1990 Aug;87(8):631-4. PMID 2395535
- [Background] de Alarcon A, Rutter MJ. Cervical slide tracheoplasty. Arch Otolaryngol Head Neck Surg. 2012 Sep;138(9):812-6. doi: 10.1001/archoto.2012.1768. PMID 22986713
- [Background] Freitag L, Darwiche K. Endoscopic treatment of tracheal stenosis. Thorac Surg Clin. 2014 Feb;24(1):27-40. doi: 10.1016/j.thorsurg.2013.10.003. PMID 24295657
- [Background] Grillo HC. Surgical treatment of postintubation tracheal injuries. J Thorac Cardiovasc Surg. 1979 Dec;78(6):860-75. PMID 502569
- [Background] Li C, Rutter MJ. Acquired tracheal stenosis: Cervical slide tracheoplasty. Semin Pediatr Surg. 2021 Jun;30(3):151058. doi: 10.1016/j.sempedsurg.2021.151058. Epub 2021 May 25. PMID 34172213
- [Background] Manning PB, Rutter MJ, Lisec A, Gupta R, Marino BS. One slide fits all: the versatility of slide tracheoplasty with cardiopulmonary bypass support for airway reconstruction in children. J Thorac Cardiovasc Surg. 2011 Jan;141(1):155-61. doi: 10.1016/j.jtcvs.2010.08.060. Epub 2010 Nov 5. PMID 21055774
- [Background] Schweiger C, Cohen AP, Rutter MJ. Tracheal and bronchial stenoses and other obstructive conditions. J Thorac Dis. 2016 Nov;8(11):3369-3378. doi: 10.21037/jtd.2016.11.74. PMID 28066618
- [Background] Smith MM, Cotton RT. Diagnosis and management of laryngotracheal stenosis. Expert Rev Respir Med. 2018 Aug;12(8):709-717. doi: 10.1080/17476348.2018.1495564. Epub 2018 Jul 12. PMID 29969925
- [Background] Tsang V, Murday A, Gillbe C, Goldstraw P. Slide tracheoplasty for congenital funnel-shaped tracheal stenosis. Ann Thorac Surg. 1989 Nov;48(5):632-5. doi: 10.1016/0003-4975(89)90777-7. PMID 2818051
- [Background] Zalzal HG, Behzadpour HK, Leonard J, Sinha P, Preciado DA. Systematic Review of Slide Tracheoplasty Outcomes. Ann Otol Rhinol Laryngol. 2023 May;132(5):558-565. doi: 10.1177/00034894221104955. Epub 2022 Jun 20. PMID 35723210